CLINICAL TRIAL: NCT04516551
Title: Anti-CD19 Donor-derived CAR-T Cells for Patients With Relapsed B Cell Malignancies After Hematopoietic Stem Cell Transplantation: a Multi-center, Uncontrolled Trial.
Brief Title: Anti-CD19 Allo-CAR-T Cells for Relapsed B Cell Malignancies After HSCT
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xinqiao Hospital of Chongqing (Other)
Collaborators: Gracell Biotechnologies (Shanghai) Co., Ltd. (Industry); First Affiliated Hospital of Zhejiang University (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); The General Hospital of Western Theater Command (Other); Chongqing University Cancer Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); Tang-Du Hospital (Other); 920th Hospital of Joint Logistics Support Force of People's Liberation Army of China (Other)
Responsible Party: Principal Investigator, Xi Zhang, MD, Chef of Hematology Department, Xinqiao Hospital of Chongqing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Anti-CD19 allo-CAR-T
Record Dates: First submitted 2020-08-13; First posted 2020-08-18 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Relapsed Adult ALL; B Cell Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD19 allo-CAR-T (Experimental): The study will employ dose level cohorts of three patients that will be treated at each level described below, based on the number of T cells to be infused using the "3 + 3" dose-escalation strategy to find MTD followed by a dose-expansion phase at determining optimal dosage.
  dosage: the number of anti CD19+CD22 CAR T cells
  -1(if needed) 1×10^6/KG
  3×10^6 /KG 6×10^6 /KG 1×10^7/KG Treatment follows a lymphodepletion, chemotherapy regimen that consists of Fludarabine (30 mg/m2 per day) and Cyclophosphamide (300mg/m2 per day) for 3 days or bendamustione (90mg/m2 per day) for two days prior to cell infusion.
  Interventions: Biological: anti-CD19 allo-CAR-T cells

INTERVENTIONS:
Biological: anti-CD19 allo-CAR-T cells — The T cells collected from haploidentical donors have been manufactured to express CAR to binding CD19 on B-cell leukemia.

SUMMARY:
The patients with relapsed B cell acute lymphoblastic leukemia (ALL) after hematopoietic stem cell transplant (HSCT) have a poor prognosis, especially for these relapsed in a short time after transplantation. Nowadays there is no effective way to salvage patients in such conditions. T cells derived from healthy matched sibling or unrelated donors have not been restrained by tumor micro-environment and retain anti-leukemia ability, which makes it serve well for patients with relapsed B-ALL. So we launched a multi-center clinical trial to proved the safety and efficacy of anti-CD19 CAR-T cells for relapsed B cell ALL.

DETAILED DESCRIPTION:
The stunning response rate of anti-CD19(cluster of differentiation antigen 19) auto-CAR(chimeric antigen receptor)-T cell therapy brings hope to patients with relapsed or refractory B-cell hematologic malignancies. However, for B-ALL patients suffered from relapse after allo-HSCT (hematopoietic stem cell transplant), the T cells derived from healthy donor seems like a better origin for CAR-T cells producing because T cells derived from healthy matched sibling or unrelated donors have not been restrained by tumor micro-environment and retain anti-leukemia ability. So after we designed a clinical trial to manifest the safety and efficacy of anti-CD19 CAR-T cells for patients with relapsed B cell ALL.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of relapsed B-cell acute lymphoblastic leukemia (B-ALL).
2. Patients have received hematologic stem cell transplantation from matching sibling donor or unrelated donor.
3. CD19-positive tumor (>20% CD19 positive blasts by flow cytometry or immunohistochemistry (tissue)）
4. Hgb ≥ 7.0 (can be transfused)
5. Life expectancy greater than 12 weeks
6. Informed consent explained to, understood by and signed by the patient/guardian. The patient/guardian is given a copy of informed consent.

Exclusion Criteria:

1. Other tumors except cured non-melanoma skin cancer, cervical cancer in situ, superficial bladder cancer, breast duct cancer in situ, or other malignant tumors with complete remission of more than 5 years)；
2. Severe mental disorders；
3. A history of genetic diseases such as Fanconi anemia, Shudder-Dale syndrome, Costman syndrome, or any other known bone marrow failure syndrome；
4. Subjects with II-IV grade acute graft versus host disease GVHD (Glucksberg Standrad) or chronic GVHD.
5. Heart disease with grade III-IV heart failure [NYHA classification], myocardial infarction, angioplasty or stenting, unstable angina or other heart diseases with prominent clinical symptoms within one year before admission；
6. Subjects with any indwelling catheter or drainage tube (such as percutaneous nephrostomy tube, bile drainage tube or pleura/peritoneum/pericardium catheter), should be excluded. (Special central venous catheter is allowed)；
7. Subjects with a history of CNS lymphoma, CSF malignant cells, or brain metastasis；
8. Subjects with a history of CNS disease,such as epilepsy, cerebral ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease involving CNS；
9. Any of the following virological ELISA results are positive: HIV antibody, HCV antibody, TPPA, HBsAg；
10. Active infection requiring systematic treatment within 2 weeks before single collection；
11. Subjects with known severe allergic reactions to cyclophosphamide or fludarabine, or diagnosed as the allergy；
12. History of autoimmune diseases (e.g. Crohn disease, rheumatoid arthritis, systemic lupus erythematosus) that cause end-organ damage or require systemic immunosuppressive medications or systemic disease modifying drugs in the past 2 years；
13. Presence of pulmonary fibrosis；
14. Subjects who have received other clinical trial treatment within 4 weeks before participating in this trial should be excluded. Or the signing date of informed consent is within 5 half-lives of the last application of another clinical trial (whichever is longer)；
15. Subjects with poor compliance due to physiological, family, social, geographical and other factors, or those unable to cooperate with the study plan or follow-up；
16. At the discretion of the investigator, there are complications requiring systemic corticosteroid therapy (≥ 5mg / day of prednisone or equivalent dose of other corticosteroids) or other immunosuppressive drugs within 6 months after this clinical research treatment；
17. The lactating woman who is reluctant to stop breastfeeding；
18. Any other condition considered unsuitable by the investigator.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2020-11-20 (Estimated); Primary Completion 2021-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
the safety of anti-CD19 allo CAR-T cells | within 4 weeks after infusion
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
the efficacy of anti-CD19 allo CAR-T cells | 4 weeks after infusion
  ratio of bone marrow blast cells

SECONDARY OUTCOMES:
The long-term efficiency | up to 2 years after infusion
  ratio of bone marrow blast cells

CONTACTS AND LOCATIONS:
Overall Officials: Xi Zhang, MD phD, Study Chair — Xinqiao Hospital of Chongqing; He Huang, MD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (1):
- Department of Hematology, Xinqiao Hospital, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Luo Y, Gao L, Liu J, Yang L, Wang L, Lai X, Gao S, Liu L, Zhao L, Ye Y, Wang M, Shen L, Cao WW, Wang D, Li W, Zhang X, Huang H. Donor-derived Anti-CD19 CAR T cells GC007g for relapsed or refractory B-cell acute lymphoblastic leukemia after allogeneic HSCT: a phase 1 trial. EClinicalMedicine. 2023 Dec 21;67:102377. doi: 10.1016/j.eclinm.2023.102377. eCollection 2024 Jan. PMID 38204488